CLINICAL TRIAL: NCT06571162
Title: A Pragmatic INitiative for LDL-C Management by a CLinical Pharmacist-Led Team Among Atherosclerotic CardiovascUlar DisEase Patients (The INCLUDE Trial)
Brief Title: A Pragmatic INitiative for LDL-C Management by a CLinical Pharmacist-Led Team Among Atherosclerotic CardiovascUlar DisEase Patients
Acronym: INCLUDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: INC 1.0
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Patients will receive usual care for their LDL-C management.
  Interventions: Other: Usual Care
- Clinical Pharmacy Team (Experimental): Patients will receive targeted care of their LDL-C through a pharmacist-driven management program.
  Interventions: Other: Clinical Pharmacy Team

INTERVENTIONS:
Other: Clinical Pharmacy Team — Patients will receive targeted care of their LDL-C through a pharmacist-driven management program.
  Arms: Clinical Pharmacy Team
Other: Usual Care — Patient will receive usual care for their LDL-C management.
  Arms: Usual Care

SUMMARY:
Patients who had an ASCVD event at an Intermountain hospital will be screened for eligibility to be randomized. Subjects who meet eligibility criteria will be randomized 1:1 to receive targeted care of their LDL-C through a pharmacist-driven management program or not. Patients may opt-out of receiving LDL-C management by the pharmacy team at any time. The purpose of this program is to increase the proportion of patients who achieve guideline-based recommendations of LDL-C levels of <70 mg/dL by increasing statin and/or LLT adherence and LDL-C testing. Data collection as part of the study will continue until the last person randomized has had 1-year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18 years of age
2. Receive follow-up care with Intermountain Health
3. Value-based patient (as defined in the EDW)
4. Documentation of an ASCVD diagnosis, by 1 of the following:

   * Coronary artery disease (Primary inpatient CAD diagnosis during index encounter; Primary inpatient MI diagnosis during index encounter; PCI during index encounter; or CABG during index encounter
   * Cerebrovascular accident (Primary inpatient ischemic stroke diagnosis during index encounter; Carotid endarterectomy during index encounter; or Carotid stent during index encounter)
   * Peripheral arterial disease (Bypass or percutaneous intervention during index encounter)

Exclusion Criteria:

1. Patient age <18 years.
2. Receipt of or expected receipt of palliative care, expected discharge to hospice, or long-term care facility (i.e., skilled nursing facility).
3. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve an LDL-C <70 mg/dL by 1-year. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Healthcare Hospitals and Clinics, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No